CLINICAL TRIAL: NCT04147052
Title: An Internet-delivered Cognitive Behavioral Intervention for Sleep Disturbance in Multiple Sclerosis
Brief Title: iSLEEPms: An Internet-Delivered Intervention for Sleep Disturbance in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00116581; K23HD086154 (NIH)
Record Dates: First submitted 2019-10-25; First posted 2019-10-31 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iSLEEPms (Experimental): Participants randomized to iSLEEPms complete a 4-week online program with telephone support, based on CBT-I.
  Interventions: Behavioral: iSLEEPms
- Treatment As Usual (No Intervention): Participants randomized to TAU continue their usual care and are encouraged to avoid starting any new sleep treatment unless deemed necessary by a health care provider.

INTERVENTIONS:
Behavioral: iSLEEPms — Participants randomized to iSLEEPms complete daily online sleep diary forms and weekly online educational modules. Modules focus on typical elements of CBT-I, adapted for individuals with MS: education about sleep in MS, sleep restriction, and stimulus control; sleep hygiene and relaxation; and cognitive restructuring around sleep and coping with MS. Sleep diaries are scored each week, and feedback is provided to participants to guide adjustments to their recommended bedtimes and wake times. Telephone support is available to provide clarification around module content.
  Arms: iSLEEPms

SUMMARY:
Sleep disturbance, especially insomnia (i.e., difficulty initiating and maintaining sleep), affects over half of people with MS. Cognitive behavioral strategies have been shown to improve sleep quantity and quality in several neurologic populations (e.g., traumatic brain injury, Parkinson's disease), and cognitive behavioral therapy for insomnia (CBT-I) is considered the first-line insomnia treatment for adults in the general population. Although cognitive behavioral interventions have historically been delivered in-person, a growing body of literature supports telephone- and internet-delivered approaches. However, more work is needed to understand the effects of internet-delivered CBT-I on patient-reported and objective outcomes.

This study is a pilot randomized controlled trial to test the preliminary effects of iSLEEPms, a CBT-I-based online intervention with telephone support for individuals with MS. After completing a baseline assessment (Week 1), 90 participants with MS will be randomized (1:1) to four weeks (Weeks 2-5) of iSLEEPms (intervention group) or treatment as usual (TAU; control group), and complete post-treatment (Week 6) and follow-up (Week 12) assessments. iSLEEPms participants will complete daily sleep diary forms and weekly online educational modules. TAU participants will continue usual care without access to the iSLEEPms materials.

The primary outcomes will be patient-reported and actigraphic measures of sleep quality and quantity. Secondary outcomes will be treatment satisfaction, adherence, and integrity (iSLEEPms group only). Exploratory outcomes will be fatigue symptoms, depression symptoms, and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and older
* MS diagnosis56 of at least 1 year duration
* Able to speak and read English
* Sleep disturbance as indicated by an ISI score of at least 11
* Willingness to commit to a 4-week intervention and 12-week follow-up assessment

Exclusion Criteria:

* Neurological disorder other than MS
* Hazardous alcohol use, as indicated by the Alcohol Use Disorders Identification Test (AUDIT-C)
* Hazardous substance use, as indicated by the Drug Abuse Screening Test (DAST-10)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Change in the Pittsburgh Sleep Quality Index (PSQI) total score | Baseline (Week 1), Post-intervention (Week 6), and Follow-up (Week 12)
  The PSQI is a 9-item participant-reported measure that assesses sleep quality. Scores range from 0 to 21 points, with higher scores indicating poorer sleep quality. Scores ≥ 5 are clinically significant.
Change in the Insomnia Severity Index (ISI) total score | Baseline (Week 1), Post-intervention (Week 6), and Follow-up (Week 12)
  The ISI is a 7-item participant-reported measure that assesses insomnia symptoms. Scores range from 0 to 28 points (each item is rated 0-4), with higher scores indicating greater insomnia. Scores ≥ 11 are clinically significant.
Change in actigraphic total sleep time (TST) | Baseline (Week 1), Post-intervention (Week 6), and Follow-up (Week 12)
  Wrist actigraphy devices objectively assess TST, in minutes. TSTs < 360 min are considered clinically significant.
Change in actigraphic sleep efficiency (SE) | Baseline (Week 1), Post-intervention (Week 6), and Follow-up (Week 12)
  Wrist actigraphy devices objectively assess SE as a % of time asleep while in bed. SEs < 85% are considered clinically significant.
Change in actigraphic sleep latency (SL) | Baseline (Week 1), Post-intervention (Week 6), and Follow-up (Week 12)
  Wrist actigraphy devices objectively assess SL, in minutes. SLs > 30 min are considered clinically significant.
Change in actigraphic wake after sleep onset (WASO) | Baseline (Week 1), Post-intervention (Week 6), and Follow-up (Week 12)
  Wrist actigraphy devices objectively assess WASO, in minutes. WASOs > 30 min are considered clinically significant.

SECONDARY OUTCOMES:
Change in the Modified Fatigue Impact Scale (MFIS) total score | Baseline (Week 1), Post-intervention (Week 6), and Follow-up (Week 12)
  The MFIS is a 21-item participant-reported measure that assesses how much fatigue impacts physical, cognitive, and psychosocial functioning. Scores range from 0 to 84 (each item is rated 0-4), with higher scores indicating a greater impact of fatigue. Scores ≥ 38 are clinically significant. The scale has three subscales (Physical, 9 items; Cognitive, 10 items; and Psychosocial, 2 items).
Change in the Beck Depression Inventory - Fast Screen (BDI-FS) total score | Baseline (Week 1), Post-intervention (Week 6), and Follow-up (Week 12)
  The BDI-FS is a 7-item participant-reported measure of depressive symptom severity. Scores range from 0 to 21 (each item rated 0-3), with higher scores indicating greater depressive symptom severity. Scores ≥ 4 are clinically significant.
Change in the MS Neuropsychological Screening Questionnaire (MSNQ) total score | Baseline (Week 1), Post-intervention (Week 6), and Follow-up (Week 12)
  The MSNQ is a 15-item participant-reported measure of subjective cognitive dysfunction. Scores range from 0 to 60 (each item rated 0-4), with higher scores indicating greater perceived cognitive dysfunction.
Change in the TestMyBrain Memorizing Words (MW) score | Baseline (Week 1), Post-intervention (Week 6), and Follow-up (Week 12)
  TestMyBrain.org is an online platform that objectively assesses cognitive dysfunction. MW is a verbal paired associates test. Participants learn and memorize 25 word pairs and are asked to recall them after a delay. Higher scores indicate better verbal memory performance.
Change in the TestMyBrain Memorizing Pictures (MP) score | Baseline (Week 1), Post-intervention (Week 6), and Follow-up (Week 12)
  TestMyBrain.org is an online platform that objectively assesses cognitive dysfunction. MP is a visual paired associates test. Participants learn and memorize 24 pictures pairs and are asked to recall them after a delay. Higher scores indicate better visual memory performance.
Change in the TestMyBrain Matching Shapes and Numbers (MSN) score | Baseline (Week 1), Post-intervention (Week 6), and Follow-up (Week 12)
  TestMyBrain.org is an online platform that objectively assesses cognitive dysfunction. MSN is a speeded digit-symbol coding task. Participants use a key provided on the screen to quickly match 9 unique symbols with their correctly paired digits as quickly as possible. Higher scores indicate faster processing speed.
Change in the TestMyBrain Fast Choices (FC) score | Baseline (Week 1), Post-intervention (Week 6), and Follow-up (Week 12)
  TestMyBrain.org is an online platform that objectively assesses cognitive dysfunction. FC is a choice reaction time test. Participants view arrows and quickly judge their direction. Higher scores indicate faster processing speed.
Treatment Satisfaction Scale (TSS) total score (iSLEEPms group only) | Post-intervention (Week 6)
  The TSS a 7-item participant-reported measure adapted from the Consumer Report Treatment Satisfaction Scale to assess satisfaction with iSLEEPms. The 7 items (each item rated 1 to 5) are averaged to calculate a total score, with higher scores indicating greater symptom improvement during the iSLEEPms program.
iSLEEPms treatment adherence (iSLEEPMS group only) | Post-intervention (Week 6)
  Treatment adherence will be assessed based on completion of each of the four weekly iSLEEPms modules, including completion of the online daily sleep diary form and weekly module. A total score will be determined based on the percentage of diary forms and weekly modules completed over four weeks.
iSLEEPms treatment integrity (iSLEEPMS group only) | Post-intervention (Weeks 6)
  Treatment integrity will be assessed based on coverage of coverage of 17 CBT-I elements, adapted from the Treatment Components Adherence Scale. A total score will be determined based on the percentage of elements covered over the four-week iSLEEPms intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Abbey J Hughes, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States